CLINICAL TRIAL: NCT01087125
Title: Abatacept Pregnancy Exposure Registry OTIS Autoimmune Diseases in Pregnancy Project: An Extension Study
Brief Title: Abatacept Pregnancy Exposure Registry
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: University of California, San Diego (Other); The Organization of Teratology Information Specialists (Other)
Responsible Party: Sponsor
Other Study IDs: IM101-121
Record Dates: First submitted 2010-03-12; First posted 2010-03-16 (Estimated); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pregnant RA patients with abatacept exposure during pregnancy
  Interventions: Drug: No Interventions

INTERVENTIONS:
Drug: No Interventions — No Interventions

SUMMARY:
The purpose of the abatacept pregnancy registry is to monitor planned and unplanned pregnancies exposed to abatacept, to evaluate the possible teratogenic effects (that is, any abnormal development) of this medication in the pregnancy outcome and to follow live born infants for one year after birth.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Currently pregnant women who agree to the conditions and requirements of the study including the interview schedule, release of medical records, and the physical examination of live born infants

Exclusion Criteria:

* Women who come in first contact with the project after prenatal diagnosis of a fetal abnormality

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2006-09-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Major structural birth defects of newborns | Throughout pregnancy and up to 1 year of life

SECONDARY OUTCOMES:
3 or more minor structural defects | at dysmorphological exam
Spontaneous abortion | throughout pregnancy
Premature delivery | throughout pregnancy
Small for gestational age | at birth
Postnatal growth deficiency | throughout pregnancy and up to 1 year of life
Postnatal serious infections, hospitalizations or malignancies | 1st year of life

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Bristol-Myers Squibb, Active, Princeton, New Jersey, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm